CLINICAL TRIAL: NCT06334913
Title: A Prospective Digital Monitoring Project Exploring Physical Activity, Patient Reported Outcome Measures and Disease Outcomes in Individuals With Myeloproliferative Neoplasms
Brief Title: A Prospective Patient Reported Outcomes and Wearables Study in Myeloproliferative Neoplasms
Status: Not yet recruiting | Type: Observational
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: IRAS 332286
Record Dates: First submitted 2024-03-13; First posted 2024-03-28 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Myeloproliferative Neoplasm
MeSH Terms: conditions — Myeloproliferative Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- MPN patients: U.K. based adult patients with MPN diagnosis.

SUMMARY:
The investigators will assess the use of a smart phone app to monitor patient reported outcomes and record biometric data in patients with myeloproliferative neoplasms.

DETAILED DESCRIPTION:
To determine whether the development of a dedicated myeloproliferative neoplasm (MPN) smartphone application is of benefit to MPN patients and shows utility for medical professionals to explore efficient disease management through retrieval of 'real-world' patient data.

1. To Track Symptoms and Provide Easy Access to Information: The core focus of the project is to enhance the quality of life for people with MPNs. The app will serve as a comprehensive toolkit to help people with MPNs proactively monitor and track their symptoms, leading to improved self-care. The App will also provide direct access to reliable, up-to-date information about MPNs, empowering users to better understand their condition and make well-informed decisions regarding their health.
2. To Contribute to Research: The app will actively contribute to MPN research by generating valuable patient-generated real-world data to inform clinical trials, treatment development, and disease understanding. Currently, most of the clinical information and data in this patient population comes from clinical trials and major academic centres. As such, there is a significant gap in recording practice and outcomes in other areas, which likely makes up a large proportion of the total patient population. The app would provide a means of monitoring patient experience, comorbidities, treatments, and outcomes, as well as highlighting unmet needs in this under-represented patient group.

A 5-year sub-study using wearables is also planned to explore symptom management and collect biometric data to assess how this correlates with symptom burden, disease specific outcomes, treatment response and quality of life. The app's data collection capabilities have the potential to revolutionize the research landscape for MPNs. By collecting large volume data from this patient group, researchers will be able to assess trends in treatment response, biomarker identification and allow optimisation of therapeutic pathways and improve design of clinical trials. This could lead to the development of new treatments being made more widely available to patients and potentially improve the lives of this patient population.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of MPN.
2. Resident in the UK
3. Aged 18 years and over.
4. Able to confidently converse in English language.
5. Access to smartphone/ mobile phone.
6. Capable of providing informed consent.
7. Physically able to stand and ambulate independently (for substudy).

Exclusion Criteria:

* Patients with a known allergic reaction to any materials in the wearable device (substudy).
* Patients who for any reason are not able to have a wearable (substudy). For example Withings ScanWatch should not be be used if the patient has an implantable electronic device such as a pacemaker or implantable cardioverter-defibrillator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: U.K. based adult patients with diagnosis of MPN.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2029-04-01 (Estimated); Study Completion 2029-04-01 (Estimated)

PRIMARY OUTCOMES:
Patient reported outcomes - Myeloproliferative Neoplasm-10 Total Symptom Score | 5 years
  The primary outcome of this study will be to characterise a baseline of healthcare data, patient reporting of symptom burden (as per MPN 10 symptom assessment form, raneg 0-100, higher scores indicative of greater symptom burden) to understand its relevance for disease-specific clinical outcomes.

SECONDARY OUTCOMES:
Healthcare adherence | 5 years
  To determine the association between patients' adherence to medication, number of hospital attendances and admissions, and data from the wearables.
Biometric data analysis - activity index | 5 years
  Wearable device tracking activity index (calories)
Biometric data analysis - sleep score | 5 years
  Wearable device tracking sleep score (0-100)
Biometric data analysis - heart rate | 5 years
  Wearable device tracking heart rate

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Harrington, MBBS PhD, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust

IPD SHARING:
Plan to Share IPD: No
No current plans to share patient data with other researchers.